CLINICAL TRIAL: NCT05595993
Title: Hypersensitivity to Phosphodiesterase 3 Inhibition in Post-Traumatic Headache: A Randomized Clinical Trial
Brief Title: Hypersensitivity to Phosphodiesterase 3 Inhibition in Post-Traumatic Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Håkan Ashina, MD, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-21067676
Record Dates: First submitted 2022-10-23; First posted 2022-10-27 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Post-Traumatic Headache
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cilostazol (Experimental): Oral administration of 200 mg cilostazol.
  Interventions: Drug: Cilostazol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol — Study participants will be allocated to receive oral administration of 200 mg cilostazol.
  Arms: Cilostazol
Drug: Placebo — Study participants will be allocated to receive oral administration of placebo.
  Arms: Placebo

SUMMARY:
To investigate whether cilostazol (phosphodiesterase 3 inhibitor) induces headache with migraine-like features in people with persistent post-traumatic headache (PTH) attributed to mild traumatic brain injury (mTBI).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years of age upon entry into screening
* History of persistent headache attributed to mild traumatic injury to the head for ≥ 12 months and in accordance with the International Classification of Headache Disorders, 3rd Edition (ICHD-3)
* ≥ 4 monthly headache days on average across the 3 months prior to screening
* Provision of informed consent prior to initiation of any study-specific activities/procedures.

Exclusion Criteria:

* > 1 mild traumatic injury to the head
* History of any primary or secondary headache disorder prior to mild traumatic injury to the head (except for infrequent episodic tension-type headache)
* History of moderate or severe injury to the head
* History of whiplash injury
* History of craniotomy
* History or evidence of any other clinically significant disorder, condition or disease (except for those outlined above) than, in the opinion of the site investigator, would pose a risk to subject safety or interfere with study evaluation, procedures or completion
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior
* Female subjects of childbearing potential with a positive pregnancy test during any study visit
* Cardiovascular disease of any kind, including cerebrovascular diseases
* Hypertension (systolic blood pressure of ≥150 mmHg and/or diastolic blood pressure of ≥100 mmHg) prior to the start of infusion on the experimental day
* Hypotension (systolic blood pressure of ≤90 mmHg and/or diastolic blood pressure of ≤50 mmHg)
* Initiation, discontinuation, or change of dosing of prophylactic medications within 2 months prior to study inclusion
* Intake of acute medications (e.g. analgesics, triptans) within 48 hours of infusion start
* Baseline headache intensity of >3 on an 11-point numeric rating scale (0 being no headache, 10 being the worst imaginable headache)
* Baseline headache with migraine-like features or self-reported baseline headache that mimics the subjects' usual headache with migraine-like features

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Migraine-Like Headache | 12 Hours
  Difference in incidence of headache with migraine-like features (0 to 12 hours) between cilostazol and placebo.

SECONDARY OUTCOMES:
Headache Intensity Scores | 12 Hours
  Difference in area under the curve (AUC) for headache intensity scores (0 to 12 hours) between cilostazol and placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Khazali HM, Christensen RH, Chaudhry BA, Melchior AG, Ashina M, Burstein R, Ashina H. Effects of PDE-3 inhibition in persistent post-traumatic headache: evidence of cAMP-dependent signaling. J Headache Pain. 2024 Apr 17;25(1):56. doi: 10.1186/s10194-024-01762-x. PMID 38627631